CLINICAL TRIAL: NCT02424149
Title: Use of Phenazopyridine for Confirmation of Ureteral Patency During Intraoperative Cystoscopy
Brief Title: Phenazopyridine for Confirmation of Ureteral Patency
Acronym: Phenazo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Katie Propst, Fellow, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HHC-2015-0008
Record Dates: First submitted 2015-04-08; First posted 2015-04-22 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Cystoscopy
MeSH Terms: interventions — Phenazopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No preoperative phenazopyridine
- Phenazopyridine (Experimental): Preoperative phenazopyridine
  Interventions: Drug: Phenazopyridine

INTERVENTIONS:
Drug: Phenazopyridine
  Other Names: Pyridium
  Arms: Phenazopyridine

SUMMARY:
In this prospective, randomized trial subjects will be randomized to receive phenazopyridine or no medication prior to pelvic reconstructive procedures that use cystoscopy to confirm ureteral patency intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Females only
* Planned surgical procedure where cystoscopy will be used to document ureteral urine flow
* Age > or = 18 years, no upper age limit
* Able and willing to consent

Exclusion Criteria:

* Planned surgical procedure where cystoscopy will not be used
* Planned surgical procedure where cystoscopy is used for a purpose other than documenting ureteral urine flow
* age <18 years
* pregnancy
* unable/unwilling to participate
* history of allergy or adverse reaction to phenazopyridine
* hepatic dysfunction
* known phenazopyridine hypersensitivity
* history of urologic surgery
* presence of ureteral stents prior to the planned surgical procedure
* concomitant suprapubic catheter placement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

REFERENCES:
- [Derived] Propst K, Tunitsky-Bitton E, O'Sullivan DM, Steinberg AC, LaSala C. Phenazopyridine for Evaluation of Ureteral Patency: A Randomized Controlled Trial. Obstet Gynecol. 2016 Aug;128(2):348-355. doi: 10.1097/AOG.0000000000001472. PMID 27399998

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenazopyridine: Preoperative oral phenazopyridine: two tablets 97.5 mg each (195 mg total)
Period: Overall Study
Arm/Group | Control | Phenazopyridine
Started | 54 | 53
Completed | 52 | 52
Not Completed | 2 | 1
Not completed — surgery cancelled | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Phenazopyridine | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (11.3) | 62.7 (9.8) | 60.19 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 52 | 104
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 52 | 52 | 104
Charlson comorbidity index [Mean (Standard Deviation); unit: scale score] — The Charlson co-morbidity index is a scale used in longitudinal studies to estimate relative risk of death from prognostic clinical covariates. Age and comorbidities are evaluated to produce a score. Minimum score is zero, there is no maximum score. Zero is predicts no risk of death based on age and comorbidities.
  scale score | 1.96 (1.5) | 2.31 (1.1) | 2.13 (1.3)
Serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.66 (0.28) | 0.63 (0.35) | 0.65 (0.32)
History or prolapse surgery [Number; unit: participants] | 7 | 12 | 19
History of urinary tract surgery [Number; unit: participants] | 6 | 9 | 15
Surgical indication: prolapse [Number; unit: participants] | 51 | 49 | 100
Surgical indication: incontinence [Number; unit: participants] | 21 | 14 | 35
Stage II or greater prolapse: anterior [Number; unit: participants] — Pelvic organ prolapse is assessed by physical exam using the Pelvic Organ Prolpase Quantification scale. The results of the exam findings are then classified into prolapse stages which range from 0 (no prolapse ) to IV (complete prolapse). Each compartment (anterior / bladder, apical / uterus / vaginal cuff, and posterior / rectum) is assigned a stage.
  participants | 46 | 46 | 92
Stage II or greater prolapse: apical [Number; unit: participants] — Pelvic organ prolapse is assessed by physical exam using the Pelvic Organ Prolpase Quantification scale. The results of the exam findings are then classified into prolapse stages which range from 0 (no prolapse ) to IV (complete prolapse). Each compartment (anterior / bladder, apical / uterus / vaginal cuff, and posterior / rectum) is assigned a stage.
  participants | 19 | 24 | 43
Stage II or greater prolapse: posterior [Number; unit: participants] — Pelvic organ prolapse is assessed by physical exam using the Pelvic Organ Prolpase Quantification scale. The results of the exam findings are then classified into prolapse stages which range from 0 (no prolapse ) to IV (complete prolapse). Each compartment (anterior / bladder, apical / uterus / vaginal cuff, and posterior / rectum) is assigned a stage.
  participants | 38 | 34 | 72
Surgical procedure performed: concomitant incontinence procedure [Number; unit: participants] — Number of participants who underwent an incontinence procedure in addition to surgery for pelvic organ prolapse
  participants | 21 | 21 | 42
Surgical procedure performed: prolapse repair without hysterectomy [Number; unit: participants] — Subjects who underwent surgical treatment of pelvic organ prolapse without a concomitant hysterectomy.
  participants | 16 | 25 | 41
Surgical procedure performed: prolapse repair with vaginal hysterectomy [Number; unit: participants] — Number of study participants who underwent surgical repair of pelvic organ prolapse with a concomitant vaginal hysterectomy.
  participants | 27 | 18 | 45
Surgical procedure performed: prolapse repair with abdominal hysterectomy [Number; unit: participants] — Number of study participants who underwent surgical repair of pelvic organ prolapse with a concomitant abdominal hysterectomy.
  participants | 1 | 1 | 2
Surgical procedure performed: prolapse repair with laparoscopic hysterectomy [Number; unit: participants] — Number of study participants who underwent surgical repair of pelvic organ prolapse with a concomitant laparoscopic hysterectomy.
  participants | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Time to Visualize Ureteral Urine Flow Intraoperatively Measured by Timing in the Operating Room
Description: Timing was performed in the operating room. Time to visualize urine efflux was started at insertion of the cystoscope into the bladder, the time was considered complete when both ureteral orifices had displayed urine efflux.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control | Phenazopyridine
Number analyzed (Participants) | 52 | 52
seconds | 160 (158) | 173 (275)
Statistical Analysis 1: Comparison: Control vs Phenazopyridine; Test type: Superiority or Other; p = 0.77, t-test, 2 sided

2. Secondary Outcome: Physician Confidence Measured by a Survey
Description: Surgeon response to the question: "I am confident that ureteral injury was ruled out in this patient" on a 5-point Likert scale where 1 = strongly disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, 5 = strongly agree
Time Frame: day of surgery (day 0)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Phenazopyridine
Number analyzed (Participants) | 52 | 52
units on a scale | 4.6 (0.49) | 4.5 (0.61)
Statistical Analysis 1: Comparison: Control vs Phenazopyridine; Test type: Superiority or Other; p = 0.73, t-test, 2 sided

3. Secondary Outcome: Additional Interventions: Measured by Use of IV Fluids, IV Lasix, IV Methylene Blue, or Ureteral Stent Placement in OR
Description: this is a composite measure and will be reported as a single value for each arm as number of additional interventions
Time Frame: day of surgery (day 0)
Measure: Number; unit: interventions
Arm/Group | Control | Phenazopyridine
Number analyzed (Participants) | 52 | 52
interventions | 4 | 3
Statistical Analysis 1: Comparison: Control vs Phenazopyridine; Test type: Superiority or Other; p = 1.0, Fisher Exact

4. Secondary Outcome: Post-operative Urethral Discomfort Measured by Pain Scales
Description: Measured prior to catheter removal using a 10 point visual analog pain scale: Zero represented no pain, Ten represented the most severe pain.
Time Frame: post operative day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Phenazopyridine
Number analyzed (Participants) | 52 | 52
units on a scale | 2.3 (2.8) | 2.1 (2.4)
Statistical Analysis 1: Comparison: Control vs Phenazopyridine; Test type: Superiority or Other; p = 0.78, t-test, 2 sided

5. Secondary Outcome: Trial of Void Results
Description: Number of subjects that failed a back-filled trial of void on the day of hospital discharge, up to 2 days after surgery.
Time Frame: Day of hospital discharge
Population: For this outcome, 96 participants were analyzed. Of the 104 participants that completed the study, only 96 underwent a trial of void.
Measure: Number; unit: participants who failed trial of void
Arm/Group | Control | Phenazopyridine
Number analyzed (Participants) | 49 | 47
participants who failed trial of void | 19 | 9
Statistical Analysis 1: Comparison: Control vs Phenazopyridine; Test type: Superiority or Other; p = 0.04, Fisher Exact

ADVERSE EVENTS:
Time Frame: From the time of surgery to 30 days post-surgery.
Arm/Group | Control | Phenazopyridine
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes